CLINICAL TRIAL: NCT04427306
Title: Biomarker Analysis of Neoadjuvant Intralesional Therapy in High Risk Early Melanoma
Brief Title: Neoadjuvant T-VEC in High Risk Early Melanoma
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: University of California, Davis (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1529612; UCDCCSO034 (Other: UC Davis Cancer Center)
Record Dates: First submitted 2020-04-07; First posted 2020-06-11 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — talimogene laherparepvec; romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (talimogene laherparepvec) (Experimental): This study all subject get the research treatment drug (talimogene laherparepvec)
  Interventions: Drug: T-Vec

INTERVENTIONS:
Drug: T-Vec — (talimogene laherparepvec) will be given prior to surgery. Standard care the patients receive the drug after sugery
  Other Names: talimogene laherparepvec; Amgen

SUMMARY:
Despite the recent notable advances in the treatment of advanced melanoma with application of growing immunotherapies, patterns of response and factors resulting in treatment failure are poorly understood. Moreover, the application of these therapeutics has been limited in the neoadjuvant setting, particularly in earlier stage disease, even though this strategy has improved tolerance and efficacy with other modalities of therapy in other cancer types.

Survival remains significantly poorer for thicker and ulcerated lesions with T3b and T4 lesions demonstrating less than 50% survival at 5 years independent of other prognostic indicators. Oncolytic viral therapies (OVT) stimulate or suppress the immune system in different ways to stop cancer cells from growing and intra-lesional OVT has demonstrated comparable efficacy and durability with greater tolerability than most effective systemic therapy. Talimogene laherparepvec (T-VEC) is the only phase III approved intra-lesional therapy in melanoma and has demonstrated significantly improved overall response rate (64%) and bystander effect (34% in uninjected lesions) in the therapeutic setting for advanced disease.

The investigators propose an open-label, Phase 2 study of talimogene laherparepvec (T-VEC), in the neoadjuvant setting for patients with high-risk, resectable primary and cutaneous melanoma prior to definitive excision. The central hypothesis of this proposal is that neoadjuvant intra-lesional therapy with T-VEC in high risk early stage melanoma will effectively treat local and subclinical distant disease by enhanced immune recognition, immunomodulation of the nodal basin, and still allow for standard of care surgery. The primary aim of this study will be to evaluate for histologic response of melanoma with secondary aim to determine changes in immune response and draining sentinel nodes as well as relationship of immune phenotype to response rate, stage and nodal burden. The investigators plan for thorough exploratory analysis of genetic and microenvironmental changes to identify actionable targets in incomplete as well as evaluation of changes in sentinel burden and subsequent rates of locoregional disease control, recurrence-free survival and overall survival in long term follow up. The investigators predict that histologic clearance of the primary tumor in the surgical specimen will be associated with improved RFS.

DETAILED DESCRIPTION:
In summary, the goal of this project is to conduct a phase II study to evaluate efficacy of Talimogene laherparepvec in the neoadjuvant setting for primary invasive melanoma in effort to improve currently poor outcomes for these tumors. This strategy has not yet been explored in early phase disease despite dramatic results seen with neoadjuvant therapeutics in other cancer types and recent clinical studies demonstrating efficacy of this approach in advanced resectable melanoma. Our ability to predict non-responder from responder to immunotherapeutic agents such as T-VEC is not yet defined and the risk of universal exposure to these systemic agents may outweigh the hypothesized benefit given the potential for immune-mediated toxicity as well as associated costs. More importantly, mechanistic dissection of pathways and molecular/immunological signatures of response and resistance offer the promise of a more rational and targeted selection of immunotherapy to maximize benefits and minimize risks. This study would be first in kind to target high earlier stage melanoma in the neoadjuvant setting with a less toxic intra-tumoral immunotherapy with key correlative endpoints regarding immune mechanisms of response.

ELIGIBILITY:
Inclusion Criteria

1. Ability to understand and willingness to sign an informed consent form.
2. Ability to adhere to the study visit schedule and other protocol requirements.
3. Men and women ≥18 years of age.
4. ECOG performance status score of 0-1 (Appendix 13.1) / Karnofsky Performance Status (KPS) performance status of 60% or greater.
5. Life expectancy ≥ 3 months.
6. Hematology parameters defined by:

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L,
   2. Platelet count ≥ 75 × 109/L, and
   3. Hemoglobin ≥ 8 g/dL (may have been transfused)
7. Blood chemistry levels defined by:

   1. Total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range
   2. AST and ALT levels ≤ 2.5 × ULN or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).
   3. INR and aPTT ≤1.5 x ULN (for patients on anticoagulation they must be receiving a stable dose for at least 1 week prior to first treatment)
   4. Creatinine clearance ≥ 30 mL/min by Cockcroft-Gault formula.
8. Subjects with active hepatitis B virus (Hep B) and with untreated hepatitis C virus (HCV) are allowed.
9. Willingness to undergo mandatory pre-treatment biopsy (unless there is adequate archival tumor specimen available) and mandatory on-treatment biopsy.
10. Female subjects who are of non-reproductive potential (i.e., post-menopausal by history - no menses for ≥1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy). Or, female subjects of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the first study drug administration.
11. Male and female subjects who agree to use highly effective method of birth control (e.g., implants, injectables, birth control pills with two hormones, intrauterine devices [IUDs], complete abstinence or sterilized partner, and female sterilization) and a barrier method (e.g., condoms, vaginal ring, sponge, etc.) during the period of therapy and for 90 days after the last dose of study drug.
12. Biopsy-proven resectable primary cutaneous melanoma > 2.0mm in depth with residual tumor or local, in-transit, or dermal oligometastatic resectable recurrence in a treatment- naïve patient not otherwise eligible for systemic therapy
13. Residual pigmented cutaneous lesion accessible to intralesional injection

Exclusion Criteria

1. Pregnant or lactating women.
2. Any psychiatric condition that would prohibit the understanding or rendering of informed consent.
3. Any significant medical condition including additional malignancies, laboratory abnormalities, or psychiatric illness that would prevent the subject from participating and adhering to study related procedures.
4. Uncontrolled concomitant disease that in the opinion of the investigator would interfere with the patient's safety or compliance on trial.
5. Severe infection that in the opinion of the investigator would interfere with patient safety or compliance on trial within 4 weeks prior to enrollment.
6. Melanoma >/= 2.0mm in depth without residual disease following biopsy
7. Previous exposure to talimogene laherparepvec or systemic therapies
8. Concurrent cancer or treatment for a concurrent cancer, except treated non-melanoma skin cancer
9. Regional or systemic metastases
10. History of evidence of symptomatic autoimmune disease requires systemic treatment (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Immunosuppressed state, including the following:

    * Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease, concurrent opportunistic infection, receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 7 days prior to enrollment.
    * Prior immunosuppressive, chemotherapy, radiotherapy (in which the field encompassed a planned injection site), biological cancer therapy, or major surgery within 28 days prior to enrollment or has not recovered to CTCAE grade 1 or better from adverse event due to cancer therapy administered more than 28 days prior to enrollment.
    * Active human immunodeficiency virus (HIV) infection
12. Active herpetic skin lesions or prior complication of herpes simplex virus-1 infection (e.g., herpetic keratitis or encephalitis).
13. Current enrollment in another clinical trial
14. Patients who are know to be sensitive to any of the products or components of T-VEC
15. Requires intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (e.g., acyclovir), other than intermittent topical use.
16. Previous treatment with talimogene laherparepvec or any other oncolytic virus.
17. Prior therapy with tumor vaccine or received live vaccine within 28 days prior to enrollment.
18. Adjuvant hormonal therapy is allowed if appropriate for planned study.
19. Prior radiotherapy in which the field does not overlap the injection sites or non- immunosuppressive targeted therapy within 14 days prior to enrollment or has not recovered to CTCAE grade 1 or better from adverse event due to cancer therapy administered more than 14 days prior to enrollment
20. History of other malignancy within the past 5 years with the following exceptions:

    * Adequately treated non melanoma skin cancer without evidence of disease at the time of enrollment
    * Adequately treated cervical carcinoma in situ without evidence of disease at the time of enrollment
    * Adequately treated breast ductal carcinoma in situ without evidence of disease at the time of enrollment
    * Prostatic intraepithelial neoplasia without evidence of prostate cancer at the time of enrollment.
21. Subjects who are unwilling to minimize exposure with his/her blood or other body fluids to individuals who are at higher risks for HSV-1 induced complications such as immunosuppressed individuals, individuals known to have HIV infection, pregnant women, or infants under the age of 3 months, during talimogene laherparepvec treatment and through 30 days after the last dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2024-05-21 (Estimated)

PRIMARY OUTCOMES:
Pathologic response | At surgery
  Clinical efficacy and biologic effect will be calculated by measuring rates of pathologic response based on assessment of immunologic response and molecular changes in residual tumors. Based on this assessment, patients will be assigned to one of the four categories described below:
  Pathologic response defined as:
  * Pathologic Complete Response (pCR, defined as 0% residual tumor)
  * Major Pathologic Response (defined as ≤10% residual tumor)
  * Partial Pathologic Response (pPR, defined as less than or equal to 50% viable tumor cells)
  * Pathologic Non-Response (pNR, defined as greater than 50% viable tumor cells)
  The analysis will be based on intent-to-treat (ITT). If a patient fails to complete treatment or disease reassessment, then he/she will be counted as a non-responder, even though the exact response is unknown.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Gaskill, MD, Principal Investigator — UC Davis Department of Surgery; Michael C Lowe, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- UC Davis Comprehensive Cancer Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/viral-therapy-in-high-risk-early-melanoma-491766/